CLINICAL TRIAL: NCT06490497
Title: Analysis of the Expectations and Needs of a Caregiver of a Glioblastoma Patient Undergoing in Oncology
Brief Title: Expectations and Needs of a Glioblastoma Caregiver
Acronym: GLOIOS
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-04
Record Dates: First submitted 2024-06-24; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Glioblastoma
Keywords: family caregiver
MeSH Terms: conditions — Glioblastoma | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregiver of a glioblastoma patient undergoing glioblastoma treated in oncology
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — individual interviews semi-directive

SUMMARY:
Cancers of the central nervous system have a poor prognosis. Glioblastoma is most common glial tumor of the central nervous system. The presence of a tumour in the brain determines the particular and specific nature of care for these patients and their families. Symptoms affect daily life and the balance of the family sphere.It's easy to imagine a difficult and disturbed family's daily routine.

Caregivers find themselves in great distress but can still benefit from support to lighten the domestic burden, and financial burden, thanks to the various recommendations of successive Cancer Plans. In fact, support for patients and their families during the illness and after is one of the key points of the programs in place. The aim of this research will be to provide food for thought in order to improve the support provided to family and friends.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of a person with glioblastoma glioblastoma undergoing oncology treatment
* Caregivers aged 18 and over

Exclusion Criteria:

- Patient's opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of a person with glioblastoma glioblastoma undergoing oncology treatment
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Difficulties and specific needs of a caregiver | Day 1
  Identify the difficulties and specific needs of a caregiver in the particular context of a person with glioblastoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No